CLINICAL TRIAL: NCT06672601
Title: The HYPA Study: Intra-abdominal Hypertension and Abdominal Compartment Syndrome in Patients Undergoing Open and Robotic Pancreatic Procedures
Brief Title: Intra-abdominal Hypertension and Abdominal Compartment Syndrome in Patients After Pancreatic Procedures.
Acronym: HYPA
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Štěpán-Ota Schütz, Surgical resident, Postgraduate student, Charles University, Czech Republic
Other Study IDs: 108/19-61/2024
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Intra Abdominal Pressure; Abdominal Compartment Syndrome; Pancreatic Surgery; Pancreatic Fistula After Pancreaticoduodenectomy; Delayed Gastric Emptying; Anastomotic Leaks; Overload Fluid
Keywords: Intra-abdominal hypertension; Compartment syndrome; Pancreatic surgery; Robotic surgery
MeSH Terms: conditions — Intra-Abdominal Hypertension; Gastroparesis; Anastomotic Leak; Edema; Compartment Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after pancreatic procedures: All patients following pancreatic procedure

SUMMARY:
This study investigates the development of intra-abdominal hypertension and compartment syndrome in patients undergoing elective pancreatic procedures. Main objective is to determine the proportion of patients after pancreatic operation who develop elevated intra-abdominal pressure and assess its association with postoperative complication rates. Another goal of the study is to compare open versus robotic pancreatic procedures regarding the occurrence of intra-abdominal hypertension and abdominal compartment syndrome.

DETAILED DESCRIPTION:
HYPA study is designed as a prospective observational study. The primary objective of this study is to assess the risk and prevalence of intra-abdominal hypertension and abdominal compartment syndrome following pancreatic procedures. The secondary objective aims to explore potential correlations between intra-abdominal hypertension and the development of postoperative complications, such as anastomotic dehiscence, postoperative pancreatic fistulas, prolonged postoperative ileus, or delayed gastric emptying. The third objective is to compare the incidence of intra-abdominal hypertension in patients undergoing robotic versus open pancreatic procedures

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18-year-old
* Indication for elective pancreatic procedure
* Written informed consent

Exclusion Criteria:

* Patients <18 years old.
* Contraindication for urinary catheter placement.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing open or robotic pancreatic procedures in our department.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Intra-abdominal hypertension and abdominal compartment syndrome | From the admission to the intensive care unit until the postoperative day 7 or until discharge from the ICU
  Prevalence of intra-abdominal hypertension and abdominal compartment syndrome in patients following pancreatic procedures.

SECONDARY OUTCOMES:
Correlation between intra-abdominal hypertension and the development of postoperative complications. | From the enrollment to the 90 days follow up period.
  The secondary objective aims to explore potential correlations between intra-abdominal hypertension and the development of postoperative complications, such as anastomotic dehiscence, postoperative pancreatic fistulas, prolonged postoperative ileus, or delayed gastric emptying.

OTHER OUTCOMES:
Incidence of Intra-abdominal hypertension in patients following robotic vs. open pancreatic procedure. | From the admission to the intensive care unit for 7 consecutive days or until discharge from the ICU.
  The tertiary objective is to compare open and robotic pancreatic procedures in terms of incidence of intra-abdominal hypertension and ACS

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Záruba, MD., Study Chair — Department of Surgery 2nd Faculty of Medicine, Charles University
Locations (1):
- Department of Surgery 2nd Faculty of Medicine, Charles University and Military University Hospital Prague, Prague, Prague 6, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie results in a publication
Supporting Information: Study Protocol

REFERENCES:
- [Background] Smit M, Koopman B, Dieperink W, Hulscher JBF, Hofker HS, van Meurs M, Zijlstra JG. Intra-abdominal hypertension and abdominal compartment syndrome in patients admitted to the ICU. Ann Intensive Care. 2020 Oct 1;10(1):130. doi: 10.1186/s13613-020-00746-9. PMID 33001288
- [Background] Reintam Blaser A, Regli A, De Keulenaer B, Kimball EJ, Starkopf L, Davis WA, Greiffenstein P, Starkopf J; Incidence, Risk Factors, and Outcomes of Intra-Abdominal (IROI) Study Investigators. Incidence, Risk Factors, and Outcomes of Intra-Abdominal Hypertension in Critically Ill Patients-A Prospective Multicenter Study (IROI Study). Crit Care Med. 2019 Apr;47(4):535-542. doi: 10.1097/CCM.0000000000003623. PMID 30608280
- [Background] Mancilla Asencio C, Berger Fleiszig Z. Intra-Abdominal Hypertension: A Systemic Complication of Severe Acute Pancreatitis. Medicina (Kaunas). 2022 Jun 10;58(6):785. doi: 10.3390/medicina58060785. PMID 35744049
- [Background] Hunter JD, Damani Z. Intra-abdominal hypertension and the abdominal compartment syndrome. Anaesthesia. 2004 Sep;59(9):899-907. doi: 10.1111/j.1365-2044.2004.03712.x. PMID 15310355
- [Background] Ball CG, Kirkpatrick AW, McBeth P. The secondary abdominal compartment syndrome: not just another post-traumatic complication. Can J Surg. 2008 Oct;51(5):399-405. PMID 18841232
- [Background] Leon M, Chavez L, Surani S. Abdominal compartment syndrome among surgical patients. World J Gastrointest Surg. 2021 Apr 27;13(4):330-339. doi: 10.4240/wjgs.v13.i4.330. PMID 33968300
- [Background] Sugrue M, Jones F, Deane SA, Bishop G, Bauman A, Hillman K. Intra-abdominal hypertension is an independent cause of postoperative renal impairment. Arch Surg. 1999 Oct;134(10):1082-5. doi: 10.1001/archsurg.134.10.1082. PMID 10522851
- [Background] Sugrue M, Buist MD, Hourihan F, Deane S, Bauman A, Hillman K. Prospective study of intra-abdominal hypertension and renal function after laparotomy. Br J Surg. 1995 Feb;82(2):235-8. doi: 10.1002/bjs.1800820234. PMID 7749700
- [Background] Gray S, Christensen M, Craft J. The gastro-renal effects of intra-abdominal hypertension: Implications for critical care nurses. Intensive Crit Care Nurs. 2018 Oct;48:69-74. doi: 10.1016/j.iccn.2018.06.001. Epub 2018 Jun 21. PMID 29937073
- [Background] De Waele JJ, De Laet I, Kirkpatrick AW, Hoste E. Intra-abdominal Hypertension and Abdominal Compartment Syndrome. Am J Kidney Dis. 2011 Jan;57(1):159-69. doi: 10.1053/j.ajkd.2010.08.034. PMID 21184922
- [Result] Kirkpatrick AW, Roberts DJ, De Waele J, Jaeschke R, Malbrain ML, De Keulenaer B, Duchesne J, Bjorck M, Leppaniemi A, Ejike JC, Sugrue M, Cheatham M, Ivatury R, Ball CG, Reintam Blaser A, Regli A, Balogh ZJ, D'Amours S, Debergh D, Kaplan M, Kimball E, Olvera C; Pediatric Guidelines Sub-Committee for the World Society of the Abdominal Compartment Syndrome. Intra-abdominal hypertension and the abdominal compartment syndrome: updated consensus definitions and clinical practice guidelines from the World Society of the Abdominal Compartment Syndrome. Intensive Care Med. 2013 Jul;39(7):1190-206. doi: 10.1007/s00134-013-2906-z. Epub 2013 May 15. PMID 23673399